CLINICAL TRIAL: NCT00938977
Title: The Obesity-Hypoventilation Syndrome: A Study Of Clinical Characteristics And Predictive Factors Of Response To Treatment With Continuous Positive Airway Pressure (CPAP) And Non-Invasive Ventilation (NIV)
Brief Title: The Obesity-hypoventilation Syndrome Study of Clinical Characteristics and Predictive Factors of Response to Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Spanish Respiratory Society (Other)
Responsible Party: Neus Salord Oleo, Hospital de la Santa Creu i Sant Pau
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HospitalSCSP
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Last update posted 2009-07-14 (Estimated); Status verified 2009-07

CONDITIONS: Obesity Hypoventilation Syndrome
Keywords: Obesity Hypoventilation syndrome; cytokines; Adipokines; continuous positive airway pressure; bilevel support ventilation; Response to continuous positive airway pressure
MeSH Terms: conditions — Obesity Hypoventilation Syndrome | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP (Active Comparator): Response to treatment before/after treatment in patients with OSAS and SOH
  Interventions: Device: CPAP
- Bilevel support ventilation (Active Comparator): Before and after effect of Bilevel support ventilation in patients with SOH without OSA
  Interventions: Device: Bilevel Support Ventilation (Non-Invasive Ventilation)

INTERVENTIONS:
Device: CPAP — Before and after effect of treatment with CPAP
  Arms: CPAP
Device: Bilevel Support Ventilation (Non-Invasive Ventilation) — before/after effect of Bilevel support ventilation
  Arms: Bilevel support ventilation

SUMMARY:
Main objective:

To describe clinical and functional characteristics of the obese hypoventilating patient; to study the relation between the obesity-hypoventilation syndrome (OHS) and the obstructive sleep apnea hypopnea syndrome (OSAHS). In the second stage of the study, to assess patient response to non-invasive mechanical ventilation (NIV) and continuous positive airway pressure (CPAP), and to identify predictors of unfavourable response to treatment.

Methodology:

* Patients: Patients with obesity degree I-III, with pCO2 awake and at rest > 45 mmHg, with no underlying pulmonary or neuromuscular lung disease; two control groups, one of non-hypoventilating obese patients and the other of obese patients with OSAHS, will also be studied over the same period.
* Design: Prospective observational study. In the first stage anthropometric, clinical, functional and metabolic data will be recorded for the obese hypoventilating patients and the two control groups (obese patients without respiratory pathology, and obese patients with OSAHS).

In the second stage patients with OHS will be divided into two subgroups: group 1: patients with polysomnography (PSG) suggestive of hypoventilation, in whom NIV treatment will be initiated; group 2: patients with PSG suggestive of OSAHS (apnea-hypopnea index >15), who will be administered CPAP. Patients will be examined one month and three months after the start of treatment. The same measurements will be carried out as at the beginning of the study, with the exception of the polysomnographic study. Nonetheless, pulse oximetry and arterial gases will be performed on waking.

Expected Results:

Patients with OHS may be characterized and differentiated from obese patients without associated respiratory pathology on the basis of clinical, functional and metabolic data.

There is a group of patients with association between OSAHS and OHS that do not respond to treatment with CPAP, and this unfavorable response can be predicted in advance.

DETAILED DESCRIPTION:
HYPOTHESIS:

Patients with OHS may be characterized and differentiated from obese patients without associated respiratory pathology on the basis of clinical, functional and metabolic data.

There is a close relation between OHS and OSAHS. It is important to define this relation more precisely because of its implications for therapy.

There is no consensus on the best ventilatory method for the treatment of OHS. In the case of an association between OSAHS and OHS the International Consensus proposes initial use of CPAP, based on empirical data. We believe that there is a group of patients that do not respond to this treatment and that this unfavorable response can be predicted in advance.

OBJECTIVES:

* To assess the clinical, functional and metabolic characteristics of the patient with obesity hypoventilation syndrome (OHS).
* To describe the frequency and characteristics of the relation between OHS and the obstructive sleep apnea hypopnea syndrome (OSAHS).
* To study the predictive factors of the response to treatment with CPAP in patients with OHS and associated OSAHS.

METHODOLOGY STUDY SETTING: Pneumology and Endocrinology Services at the Hospital de la Santa Creu i Sant Pau. Hospitalization Unit, Sleep Clinic and Pulmonary Function Laboratory.

PATIENTS: Patients from a conventional hospitalization unit, semi-critical care unit, Endocrinology Clinic, Pneumology Clinic and/or Sleep Clinic meeting the following criteria:

* Obesity degree I-III (Body mass index, BMI >30 Kg/m2)
* Stable daytime PCO2 >45 mmHg.
* Age < 75 years
* Absence of other parenchymal, respiratory or neuromuscular diseases, diseases of the chest wall which may occur concomitantly with hypoventilation.
* Absence of exclusion criteria.

Exclusion criteria:

* Cognitive disorders that interfere with the administration of the clinical questionnaires.
* Grave comorbidity.
* FEV1/FVC ratio < 65% in the forced spirometry.

CONTROL GROUP:

In parallel, two control groups will be studied:

* A group of obese patients with similar age, sex and BMI. Subjects will be included if their pCO2< 45 mmHg and if the nocturnal pulse oximetry and specific clinical questionnaire are not suggestive of OSAHS.
* A group of obese patients with the same characteristics as above, but with diagnosis of OSAHS by polysomnograph or polygraph study.

STUDY VARIABLES:

* Anthropometric and socio-demographic data: age, sex, weight, height, BMI, waist circumference (above the iliac crest), neck diameter. Age of onset of obesity and length of period of obesity.
* General clinical questionnaire: family history, history of episodes of acute respiratory insufficiency, cardiovascular risk factors and comorbidity.
* Subjective assessment of degree of sleepiness: analysed using the Epworth scale (MW Johns, Sleep 1991, 14;540).
* Degree of sleepiness according to the definition of the American Thoracic Society: classification in four categories: absent, mild, moderate and grave.
* Study of respiratory function:
* Forced spirometry and inspirometry. Maximum F/V loop performed with datapir 500 spirometer (SIBEL, Barcelona), in accordance with the norms and reference values of the SEPAR (Roca et al. Respir Med. 1998 Mar;92(3):401-7.
* Static lung volumes. Measured in accordance with the norms and reference values of the SEPAR (Roca et al. Respir Med 1998 Mar;92(3):454-60.
* Arterial gases at rest. Maximum respiratory pressures (PIMAX, PEMAX): using the method described by Morales P. et al (Arch de Bronconeumol 1998; 34: 142-151)
* Conventional polysomnography (PSG). PSG will be performed during an entire night using Siesta, Compumedics equipment, recording two channels of the electroencephalogram, electrooculogram, electromyogram of chin muscles, hemoglobin saturation by pulse oximetry, oro-nasal flow by means of thermistor, thoracic and abdominal movements, electrocardiogram, anterior tibial electromyogram and body position. Sleep staging will be manual, following the classical criteria of Rechschaffen & Kales. The minimum recording time will be 6 hours, and the total time of minimal sleep will be 3 hours.

Definition of apnea: absence of flow for at least 10 s. Definition de hypopnea: any reduction in the flow of at least 10 s, accompanied by a desaturation (a noticeable fall in saturation with rapid recovery) and/or transitory waking or arousal (defined according to the ASDA criteria: Sleep, 1992; 15: 173-184). Definition of hypoventilation: Prolonged periods of arterial desaturation not preceded by episodes of respiratory events.

The following data will be recorded: number of apnea/hypopnea episodes per hour (IAH), percentage of time in apnea and/or hypopnea, number of arousals/hour, sleep efficiency (total sleep time /length of recording), percentage of time in phases 1, 2, 3-4 and REM, initial saturation, mean saturation, minimal saturation, time with saturation below 90% (CT90).

* Radioimmunoassay determination of the level of leptin in serum, determination of baseline insulinemia, determination of TSH, lipids study (triglycerides, cholesterol (total cholesterol, HDL, VDL, LDL, Apo-B)
* Adjustment of the optimal level of CPAP: after a second conventional polysomnography study, the optimal level of CPAP will be adjusted in the patients who present an IAH >15 on conventional polysomnography.
* Questionnaire on compliance with, and side effects of, CPAP/VNI treatment.

PROCEDURE:

First phase: All patients from the semicritical unit, conventional ward, pneumology outpatient service and the Sleep Clinic who meet the entry requirements will be included. Patients recruited in acute phase will be placed in the pre-inclusion group and will be definitively included in the study once their condition has been stable for 6 weeks.

A sample of obese control patients (BMI>30 Kg/m2 and pCO2 below 45 mmHg), who do not present the exclusion criteria described above, will be recruited.

RECRUITMENT PERIOD: At the start of the recruitment period the patients will be informed of the nature of the study and will be asked to give written consent to participate. Then, the data on the study variables will be compiled: anthropometric and sociodemographic data, general and specific clinical questionnaire, degree of sleepiness, study of respiratory function, leptin, baseline insulinemia, and conventional polysomnography.

In the control patients polysomnography will be performed if they present clinical symptoms suggestive of OSAHS or hypoventilation and/or CT 90 > 1% on the nocturnal ambulatory oximetry (L. Hernandez Plaza et al. Eur Resp J 1996; 9:74S).

Second phase: After the polysomnographic study two population groups will be defined: Group 1: OHS patients: polysomnographic study suggestive of hypoventilation without associated OSAHS.

Group 2: Patients with OHS and OSAHS: polysomnographic study suggestive of hypoventilation associated with OSAHS: IAH>15, with a predominance of obstructive events (>50%).

Patients in group 1 (patients with OHS) will begin NIV treatment, using a BIPAP ventilator in Spont/timed mode (RF 12) and nasal masks. The parameters of the respirator will be adjusted during a nap; expiratory pressure (EPAP) will be at least 4 cm H2O and inspiratory pressure 10-20 cm H2O, depending on the patient's tolerance. Oxygen will be added until a continuous saturation of between 93-95% is obtained, and a gas sample will be taken on waking.

In patients in group 2 a CPAP titration study will be carried out. The pressure will be adjusted on the basis of a new polysomnographic study. Once the optimum pressure is established, a nocturnal pulse oximetry will be performed and arterial gases assessed on waking.

Treatment response will be considered inadequate and the CPAP treatment discontinued during the night of titration if:

* Patients' tolerance of treatment is poor.
* There is no correction of obstructive events and/or episodes of hypoventilation.

In this case NIV treatment will be initiated, following the procedure described in group 1.

FOLLOW-UP:

T1: One month after the beginning of treatment with CPAP/VNI. Patients will be administered a questionnaire assessing clinical symptoms, compliance and side effects of treatment, physical examination, and arterial gases at rest.

T3: After three months the same measurements will be carried out as at the beginning of the study, with the exception of the polysomnographic study. Nonetheless, pulse oximetry and arterial gases will be performed on waking, using the treatment method assigned.

All patients who present clinical or gasometric deterioration during follow-up requiring a change of treatment will be excluded.

STATISTICAL ANALYSIS:

Initially, univariate analysis will be performed on the variables recorded in the patients and control groups. The results of the categorical variables will be expressed in percentages and those of the continuous variables as means + standard deviation, as median or range depending on the form of their distribution. Groups will be compared with the chi-squared text or through means comparison as required. Subsequently, the variables for which relations are found and those considered clinically important will be included in the multivariate logistical regression model in order to determine a predictive model of the presence of hypercapnia.

In the second stage of the study, over a 12-week period, the baseline and final scores of the variables will be compared using the most suitable statistical test. A p value < 0.05 will be considered significant.

The same analysis will be conducted to evaluate the relation between the different variables and the presence of OSAHS.

ELIGIBILITY:
Inclusion Criteria:

* Obesity degree I-III (Body mass index, BMI >30 Kg/m2)
* Stable daytime PCO2 >45 mmHg.
* Age < 75 years
* Absence of other parenchymal, respiratory or neuromuscular diseases, diseases of the chest wall which may occur concomitantly with hypoventilation.
* Absence of exclusion criteria.

Exclusion Criteria:

* Cognitive disorders that interfere with the administration of the clinical questionnaires.
* Severe comorbidity.
* FEV1/FVC ratio < 65% in the forced spirometry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2003-06; Primary Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neus Salord, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Mercedes Mayos, MD, Study Chair — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Salord N, Mayos M, Miralda RM, Farre A, Carreras M, Sust R, Masuet-Aumatell C, Rodriguez J, Perez A. Continuous positive airway pressure in clinically stable patients with mild-to-moderate obesity hypoventilation syndrome and obstructive sleep apnoea. Respirology. 2013 Oct;18(7):1135-42. doi: 10.1111/resp.12131. PMID 23714281